CLINICAL TRIAL: NCT04787627
Title: Clinical Investigation (Beta) of Power Knee
Brief Title: Clinical Investigation (Beta) of Power Knee Mainstream - Dynamic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Medical Center Orthotics and Prosthetics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIP2019050213
Record Dates: First submitted 2020-12-29; First posted 2021-03-08 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prosthesis User; Amputation

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized two group cross-over study, within subject comparison.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Power Knee before prescribed prosthesis (Experimental): Power Knee, the investigational device is fitted on subjects and they use it as their primary prosthesis for 2 weeks before coming in for data collection on the device. After being on the investigational device for 2 weeks subjects go back on their prescribed prosthesis for 2 weeks and comparator data is collected.
  Interventions: Device: Power Knee
- Power Knee after Prescribed prosthesis (Experimental): Subjects start the study by using their prescribed prosthesis for 2 weeks, then they come in for data collection of comparator data, in that same visit they are fitted with the investigational device and wear that for 2 weeks before coming in for data collection on that device.
  Interventions: Device: Power Knee

INTERVENTIONS:
Device: Power Knee — Powered microprocessor controlled prosthetic knee

SUMMARY:
Prospective two group cross over investigation, comparing the investigational device (Power Knee, a powered microprocessor controlled prosthetic knee) and subjects prescribed microprocessor prosthetic knee (MPK).

The primary objective was to evaluate the efficacy of the investigational device in reducing exertion during walking compared to passive MPKs. Additionally to evaluate the efficacy of the investigational device in the short and long term compared to passive MPKs and previous versions of the Power Knee, during daily living activities i.e. walking on level ground, in stairs and inclines, rising from and sitting down to a chair as well as performance of gait functions and ease of set up for average to highly active transfemoral/knee disarticulation amputees and Certified Prosthetists/Orthotists (CPOs).

DETAILED DESCRIPTION:
This is a prospective two group cross-over study, within subject comparison. 3 study visits are planned for amputee subjects, with approximately 2-3 weeks between visits, and an optional fourth visit 8-12 weeks after the third visit. During the first visit subjects will be check for inclusion/exclusion, consented and randomly assigned into two groups and Group 1 (transitioning to the investigational device) will perform functional tests and answer questionnaires on the performance of their current prosthesis to provide baseline information. The Group 1 subjects will be fitted and trained on the investigational device and a recommended prosthetic foot which they will use as their prescribed prosthesis for 2-3 weeks until the second visit, the other half will stay on their prescribed prosthesis until the second visit.

During the second visit the subjects of Group 1 will perform the same functional tests as in the first visit on the investigational device and answer questionnaires on the performance of the investigational device, and then return to their prescribed prosthesis. The Group 2 will perform the same tests/questionnaires on their prescribed prosthesis and then be fitted and trained on the investigational device and use it as their usual prosthesis for 2-3 weeks.

During the third visit all subject will repeat the tests and questionnaires on the prosthesis they are fitted with (Group1 on the prescribed and Group 2 on the investigational device). Subjects will have the option to use the investigational device for an additional 8-12 weeks, those who choose that will be fitted with the investigational device or will stay on it, depending in which they are in at this point. They will be booked for the fourth visit; they will be contacted via telephone 4-5 weeks later and asked to provide feedback on their experience with the device so far. Those that choose not to keep using the investigational device will be returned to their prescribed prosthesis.

During the fourth visit subjects will answer the same questionnaires and perform the same functional tests as the other visits. Data will be collected from the knee on activity. They will then be fitted back to their prescribed prosthesis.

End of study. CPO (Certified Prosthetist Orthotist) subjects will answer a questionnaire on the ease of setup of the investigational device and provide feedback on the ease of setup of gait functions.

Statistical considerations:

Outcomes at each timepoint were visually inspected for normality using histograms and qq-plots, as well as a Shapiro-Wilk Normality Test. If the data were deemed to be normal the hypotheses were tested using a two-tailed, paired, student's t-test. Non-normal data was tested using the Wilcoxon signed-rank test.

ELIGIBILITY:
Inclusion Criteria:

* 50Kg< body weight < 116Kg
* K3-K4 amputees with unilateral transfemoral amputation or Knee disarticulation
* Allows for 37mm knee center height to dome of pyramid alignment
* Currently using a MPK or Power Knee
* Older than 18 years old
* No socket issues/changes in the last 6 weeks and no socket changes expected during the duration of the study period.
* Comfortable and stable socket fit
* Willing and able to participate in the study and follow the protocol

Exclusion Criteria:

* 50Kg> body weight > 116Kg
* Bilateral amputees
* Users with socket problems
* Users with co-morbidities in the contra-lateral limb, which affect their functional mobility
* Younger than 18 years old
* Users with stump pain
* Users with cognitive impairment
* Users not involved in other clinical tests and/or receiving treatment that the testing might affect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Fothergill, CPO, Principal Investigator — Medical Center Orthotics and Prosthetics (MCOP) Silver Spring; John Warren, CPO, Principal Investigator — Medical Center Orthotics and Prosthetics (MCOP) Boston
Locations (2):
- United States (2):
  - Medical Center Orthotics and Prosthetics, Silver Spring, Maryland
  - Medical Center Orthotics and Prosthetics, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Power Knee Before Prescribed Prosthesis | Power Knee After Prescribed Prosthesis
Started | 9 | 8
Completed | 4 | 7
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Excluded | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Combined Crossover Evaluation Group: For the analysis, data from both arms were combined.
  In Group 1, participants initially used the investigational device, with the second visit corresponding to its evaluation after two weeks of use, and evaluated their prescribed device during the third visit, also after two weeks of use.
  In Group 2, participants started with the prescribed device, evaluating it during the second visit after two weeks of use, and switched to the investigational device for the evaluation during the third visit, again after two weeks of use.
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 52 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Amputation level Transfemoral [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Borg Category Rating Scale Before and After 6MWT at 2 Weeks
Description: Mean difference in perceived exertion on the Borg rating scale of perceived exertion before and after 6 minute walk test (6MWT) (see outcome 2) with investigational device (Power Knee) compared to comparator (prescribed device). Subjects are asked how exerted they feel on a scale of 0-10 (0 indicating no exertion and 10 indicating the most exertion) at rest before they carry out the 6MWT, and after carrying out the 6MWT, the difference is recorded.
  The Borg Category Rating 10 scale (CR10) is a validated measure of perceived exertion.
Time Frame: At baseline, after 2 weeks of either using the Power knee or their own prescription prosthesis, and at the fourth follow-up (at approximately weeks 22-16)
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Combined Crossover Evaluation Group "Combined Crossover Evaluation Group": For the analysis, data from both arms were combined.
  In Group 1, participants initially used the investigational device, with the second visit corresponding to its evaluation after two weeks of use, and evaluated their prescribed device during the third visit, also after two weeks of use.
  In Group 2, participants started with the prescribed device, evaluating it during the second visit after two weeks of use, and switched to the investigational device for the evaluation during the third visit, again after two weeks of use.
- Subset of 6 Subjects Who Opted for a Prolonged Follow up Period: Out of the eleven subjects who completed the trial, six of them opted in for an optional extended follow up period on the investigational device, and fourth visit. No subjects were lost to follow up.
Arm/Group | Combined Crossover Evaluation Group "Combined Crossover Evaluation Group" | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks : Power Knee | 3.4 (2.5) | 2.8 (1.7)
  After 2 weeks : Prescribed knee | 3.1 (1.5) | 2.5 (0.9)
  At Baseline: Prescribed knee | 3.4 (1.6) | 3.3 (1.4)
  After a prolonged follow up period : Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period : Power Knee |  | 3.2 (0.7)

2. Primary Outcome: Average Distance Walked in 6 Minute Walk Test
Description: Average distance walked in 6MWT with investigational device (Power Knee) compared to comparator (prescribed device) User walk for 6 minutes in their self selected walking speed on a 30 meter track.
  Shorter time indicates better mobility performance.
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
meters
  After 2 weeks: Power Knee | 381.7 (137.1) | 402.5 (151.5)
  After 2 weeks: Prescribed knee | 377.2 (108.6) | 390.7 (136.0)
  At Baseline : Prescribed knee | 369.2 (113.4) | 381.5 (140.3)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 393.1 (112.1)

3. Secondary Outcome: Total Score of Prosthesis Mobility Questionnaire (PMQ) Questions 9 and 10
Description: Support in sit to stand and stand to sit evaluation:
  Total score (minimum score 0 - maximum score 8) of Prosthetic Mobility Questionnaire (PMQ) questions 9 and 10 with investigational device (Power Knee) compared to comparator (prescribed knee):
  PMQ : Over the past 2 weeks, please rate your ability in the following activities when using your prosthesis (0=no ability, 4=fully able):
  * Question 9. To sit down and get up from a chair with a high seat (e.g. a dining chair, an office chair)
  * Question 10. To sit down and get up from a low, soft chair (e.g. a deep sofa) A higher total score on these PMQ items indicates a better outcome as it reflects greater functional ability, independence, and overall quality of life for individuals using a prosthesis.
  The total score is obtained by summing the scores from questions 9 and 10.
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 6.8 (1.3) | 7.2 (1.0)
  After 2 weeks: Prescribed knee | 5.8 (1.9) | 5.7 (2.1)
  At baseline: Prescribed knee | 5.6 (2.2) | 6.0 (1.4)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 6.3 (1.2)

4. Secondary Outcome: Average Score of Modified Prosthesis Evaluation Questionnaire (PEQ) Question 14F
Description: Average score with investigational device (Power Knee) compared to comparator (prescribed device) of modified PEQ Question 14F
  Modified PEQ question 14F :
  Over the past 2 weeks, please rate your ability in the following activities when using your prosthesis :
  • Question 14F. Your safety when walking down a steep hill using the prosthesis The scale used is a Likert Scale 1-10 (1 indicating low rating of safety and 10 indicating a high rating of safety).
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks : Power Knee | 7.9 (1.6) | 8.3 (1.2)
  After 2 weeks : Prescribed knee | 7.1 (2.4) | 6.8 (2.0)
  At Baseline: Prescribed knee | 7.3 (2.0) | 6.8 (1.8)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 6.7 (3.4)

5. Secondary Outcome: Average Score of Modified Prosthesis Evaluation Questionnaire (PEQ) Question 13D
Description: Average score with investigational device (Power Knee) compared to comparator (prescribed device) of modified PEQ Question 13D
  Over the past 2 weeks, please rate your ability in the following activities when using your prosthesis :
  • Question 13D.Your safety when walking downstairs using the prosthesis The scale used is a Likert Scale 1-10 (1 indicating low rating of safety and 10 indicating a high rating of safety).
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 9.2 (0.8) | 9.5 (0.6)
  After 2 weeks: Prescribed Knee | 7.8 (2.0) | 7.2 (2.2)
  At baseline: Prescribed Knee | 7.7 (1.9) | 7.7 (1.6)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 8.2 (4.0)

6. Secondary Outcome: Satisfaction With Walking Speed
Description: Proportion of subjects reporting satisfaction with walking speed on investigational device
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Number; unit: percentage of participants
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
percentage of participants | 100 | 100

7. Secondary Outcome: Prosthetic Limb Users Survey of Mobility (PLUS-M) T-score
Description: Ability to ambulate over typical environmental obstacles measured by the Prosthetic Limb Users Survey of Mobility (PLUS-M), T-score with Power Knee compared to comparator (prescribed device).
  The Prosthetic Limb Users Survey of Mobility™ is a self-report instrument for measuring mobility of adults with lower limb amputation.
  Scoring a PLUS-M short form produces a T-score. To find the T-score, the scores must be summed for all responses on the short form (creating a raw score). Then the raw score needs to be used to determine the T-score in the conversation table provided with the PLUS-M questionnaire.
  The T-score is a standardized score with a mean of 50 and a standard deviation of 10. A higher T-score indicates a higher level of mobility. The highest possible T-score is 71.4 and the lowest one is 21.8.
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 57.2 (7.9) | 57.9 (6.2)
  After 2 weeks: Prescribed Knee | 51.7 (10.2) | 51.9 (10.1)
  At Baseline: Prescribed Knee | 53.1 (9.1) | 54.1 (8.3)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 56.3 (6.3)

8. Secondary Outcome: Average Score of Modified Prosthesis Evaluation Questionnaire (PEQ) Question 13A
Description: Average score with investigational device (Power Knee) compared to comparator (prescribed device) of modified PEQ Question 13A
  Over the past 2 weeks, please rate your ability in the following activities when using your prosthesis :
  • Question 13A. Your safety (during stance phase) when walking with your prosthesis (prescribed device) /test prosthesis (Power Knee)? The scale used is a Likert Scale 1-10 (1 indicating low rating of safety and 10 indicating a high rating of safety).
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 8.4 (2.1) | 9.0 (1.6)
  After 2 weeks: Prescribed Knee | 8.5 (1.7) | 8.3 (1.9)
  At Baseline: Prescribed Knee | 8.6 (1.4) | 8.7 (1.2)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 8.0 (4.0)

9. Secondary Outcome: Average Score of Prosthesis Evaluation Questionnaire (PEQ) Question 1D
Description: Average score with investigational device (Power Knee) compared to comparator (prescribed device) of modified PEQ Question 1D
  Over the past 2 weeks, please rate your ability in the following activities when using your prosthesis :
  • Question 1D. Your comfort while standing when using your prosthesis/test prosthesis? The scale used is a Likert Scale 1-10 (1 indicating low rating of safety and 10 indicating a high rating of safety).
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 9.0 (2.1) | 9.5 (0.8)
  After 2 weeks: Prescribed Knee | 8.5 (1.2) | 8.0 (1.4)
  At Baseline: Prescribed Knee | 8.6 (1.1) | 8.3 (1.4)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 7.7 (3.4)

10. Secondary Outcome: Average Score Regarding the Ease of Setup
Description: Self reported ease of setup of investigational device compared to state of the art microprocessor knees (SOTA MPKs) and previous version of the investigational device.
  Average score with investigational device (Power Knee) compared to comparator (previous version of Power Knee) and compared to state of the art microprocessor knees (SOTA MPKs) The scale used is a Likert Scale 1-10 (1 indicating low rating and 10 indicating a high rating).
Time Frame: Immediately after the intervention (fitting of the investigational device)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Certified Prosthetist Orthotists: CPO subjects will answer a questionnaire on the ease of setup of the investigational device compared to previous version of the Power Knee and provide feedback on the ease of setup of gait functions.
Arm/Group | Certified Prosthetist Orthotists
Number analyzed (Participants) | 6
score on a scale
  Power Knee | 9.0 (1.3)
  Previous version of Power Knee | 6.5 (3.3)
  SOTA MPKs | 8.6 (1.2)

11. Secondary Outcome: Proportion of Participants With Average Score Over 5 on Questions 3K and 3L of the Prosthesis Evaluation Questionnaire (PEQ) With the Investigational Device
Description: Proportion of participants with Average score with investigational device of PEQ questions 3K and 3L over 5
  PEQ- Questions 3K, 3L:
  * Question 3K: Over the past two weeks, rate how often the test prosthesis made squeaking, clicking, or belching sounds The scale used is a Likert Scale 1-10 (1 indicating low frequency of prosthesis making sounds and 10 indicating a high frequency of the prosthesis making sounds).
  * Question 3L: 3L: If it made any sounds in the past four weeks, rate how bothersome these sounds were to you. - Or check It made no sounds The scale used is a Likert Scale 1-10 (1 indicating low frequency of prosthesis making sounds and 10 indicating a high frequency of the prosthesis making sounds).
  Support question (yes/no) "Would the noise from the test device prevent you from preferring it as your usual prosthesis?"
Time Frame: After 2 weeks of either using the Power Knee or their own prescribed knee
Measure: Number; unit: percentage of participants
Arm/Group | Combined Crossover Evaluation Group
Number analyzed (Participants) | 11
percentage of participants | 72

12. Secondary Outcome: Total Score of Prosthesis Mobility Questionnaire (PMQ) Questions 1 and 3-6:
Description: Total score of PMQ questions 1,3-6 (minimum score 0 - maximum score 20):
  PMQ (Questions 1 and 3-6):
  Over the past 2 weeks, please rate your ability in the following activities when using your prosthesis:
  * Question 1: To walk indoors
  * Question 3: To walk upstairs
  * Question 4: To walk downstairs
  * Question 5: To walk up a steep hill
  * Question 6: To walk down a steep hill The scale used is a Likert scale 0-4 (0= Unable or hardly able at all, 1= High difficulty, 2= Moderate Difficulty, 3= Little difficulty, 4= No problems or almost fully able).
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 15.6 (3.4) | 16.7 (2.4)
  After 2 weeks: Prescribed Knee | 14.2 (4.3) | 13.3 (4.2)
  At Baseline: Prescribed Knee | 13.8 (4.2) | 13.2 (3.4)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 15.8 (2.9)

13. Secondary Outcome: Time Required to Complete the L-test
Description: The L-Test of Functional Mobility consists of a series of movements designed to assess an individual's physical function and dynamic balance. The test involves the participant starting from a seated position, standing up, walking a short distance, turning, walking back, and returning to the seated position. The course typically forms an "L" shape, which includes two turns, and the total distance covered is longer than that of similar tests like the Timed Up and Go (TUG) test. The outcome measure is the time taken to complete these movements, providing an objective evaluation of the participant's functional mobility. There is no fixed minimum or maximum; lower times indicate better performance (i.e., faster completion reflects greater mobility).
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Combined Crossover Evaluation Group | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
seconds
  After 2 weeks: Power Knee | 26.3 (11.9) | 25.2 (12.6)
  After 2 weeks: Prescribed Knee | 24.2 (9.4) | 23.8 (11.7)
  At Baseline: Prescribed Knee | 23.7 (8.2) | 23.0 (10.0)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 24.1 (10.8)

14. Secondary Outcome: Average Prosthetic Mobility Questionnaire (PMQ) Total Score
Description: Average Prosthetic Mobility Questionnaire (PMQ) total score (minimum score 0 - maximum score 48) with investigational device (Power Knee) compared to comparator (prescribed device).
  The Prosthetic Mobility Questionnaire is a tool for assessing mobility in people with lower-limb amputation, higher score indicates better mobility performance.
Time Frame: as for outcome 1
Population: Only 6 out of the 11 subjects decided to do a prolonged follow up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Power Knee: FU on Power Knee for 2 weeks
Arm/Group | Power Knee | Subset of 6 Subjects Who Opted for a Prolonged Follow up Period
Number analyzed (Participants) | 11 | 6
score on a scale
  After 2 weeks: Power Knee | 35.5 (7.4) | 37.3 (4.5)
  After 2 weeks: Prescribed Knee | 31.2 (10.3) | 29.8 (9.8)
  At Baseline: Prescribed Knee | 31.5 (9.8) | 31.5 (7.2)
  After a prolonged follow up period: Power Knee: number analyzed (Participants) | 0 | 6
  After a prolonged follow up period: Power Knee |  | 35.2 (5.6)

15. Secondary Outcome: Occurrence of Side Effects That Could be Directly Related to Using the Power Knee
Description: Evaluating the occurrence of side effects associated with the Power Knee entails systematically documenting and analyzing any adverse effects experienced by users throughout the 2 weeks of use.
Time Frame: After 2 weeks of using the Power Knee
Population: For this outcome measure, side effects were assessed only after 2 weeks of Power Knee use. Although the study followed a crossover design, the timing or order in which participants used each device did not affect the evaluation of side effects. No side effect data were collected for the prescribed prosthesis; therefore, results are reported solely for the Power Knee group, reflecting all participants who completed the 2-week evaluation. Reporting by arm is not applicable for this outcome.
Measure: Number; unit: side effect
Groups:
- Power Knee Group: Participants who completed 2 weeks of use with the Power Knee, regardless of the order in which they used the devices during the crossover study.
Arm/Group | Power Knee Group
Number analyzed (Participants) | 11
side effect | 0

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- Power Knee Group: Participants during periods of Power Knee use
- Prescribed Prosthesis Group: Participants during periods of prescribed prosthesis use
Arm/Group | Power Knee Group | Prescribed Prosthesis Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 3/17 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Power Knee Group (N=17) | Prescribed Prosthesis Group (N=17)
Fall (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to Covid restrictions replacement of drop-outs was not attempted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT04787627/Prot_SAP_002.pdf